CLINICAL TRIAL: NCT07366658
Title: A Study to Explore the Safety, Tolerability, and Preliminary Efficacy of NEUK203-13 Injection in Patients With Neuroendocrine Tumors Who Have Failed Systemic Therapy
Brief Title: Safety, Tolerability and Preliminary Efficacy of NEUK203-13 in Refractory Neuroendocrine Tumor Patients
Acronym: NEUK203-13
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Neukio Biotherapeutics (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEUK203-13-IIT-01
Record Dates: First submitted 2026-01-04; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: SCLC, Extensive Stage; Neuroendocrine Tumors
Keywords: Car-NK cells; iPSC
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Biological Products; Engineering

STUDY DESIGN:
Intervention Model Description: Two dose groups are preset. For the first subject in the initial dose group, NEUK203-13 Injection is administered intravenously at a dose of 2×10⁹ cells, once every 3 days (Q3D) for a total of 3 consecutive doses. The Safety Monitoring Committee (SMC) may decide to proceed to the second dose group based on the available safety/tolerability data and pharmacokinetic/biomarker data. For subjects in the second dose group, NEUK203-13 Injection is administered intravenously at a dose of 4×10⁹ cells, once every 3 days (Q3D) for a total of 3 consecutive doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous infusion of NEUKIO203-13 was administered following lymphodepletion (Experimental): Intravenous infusion of NEUKIO203-13 was administered following lymphodepletion with cyclophosphamide combined with fludarabine.
  Interventions: Biological: Biological/Vaccine: NK Cell Therapy Product Derived from Induced Pluripotent Stem Cells (iPSCs) Engineered with Anti-DLL3 CAR Construct, Followed by Differentiation and Expansion

INTERVENTIONS:
Biological: Biological/Vaccine: NK Cell Therapy Product Derived from Induced Pluripotent Stem Cells (iPSCs) Engineered with Anti-DLL3 CAR Construct, Followed by Differentiation and Expansion — Intravenous infusion of NEUKIO203-13 d1,d4,d7 and IL-2 6 mIU d1,d4,d7 and d10 was administered following lymphodepletion with cyclophosphamide combined with fludarabine.

SUMMARY:
This is a Phase I clinical trial being conducted in humans for the first time, aiming to evaluate a novel cell therapy called NEUK203-13 Injection for the treatment of patients with advanced small cell lung cancer (SCLC) who have failed systematic therapy or late stage neuroendocrine tumors(NETs). The primary goal of the study is to determine the safety and tolerability of this new therapy and to preliminarily observe its anti-tumor effects.

NEUK203-13 Injection is an "off-the-shelf" CAR-NK cell therapy developed based on induced pluripotent stem cell (iPSC) technology, targeting the DLL3 protein highly expressed in SCLC or other neuroendocrine tumors(NETs) .

Primary Objective Primary Endpoint aims to evaluate safety and tolerability Secondary Endpoints aim to preliminarily observe efficacy and investigate the pharmacokinetics of the drug in the body.

Two pre-set dose levels are planned, with an enrollment of 7-9 patients. Treatment Regimen

1. Lymphodepletion Conditioning: Chemotherapy (Cyclophosphamide + Fludarabine) before cell infusion to clear lymphocytes in the body.
2. Cell Infusion: NEUK203-13 is administered via intravenous infusion, d1，d4 and d7 for three doses.
3. Supportive Medication: Concurrent use of IL-2 (Interleukin-2) d1, d4, d7 and d10 to support NK cell persistence.

Target Patient Population Patients with advanced SCLC who have progressed after prior platinum-based chemotherapy or late stage neuroendocrine tumors(NETs) and have a relatively good performance status.

Key Monitoring Focus Close monitoring of risks specific to cell therapy, such as Cytokine Release Syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS).

In short, this study represents the first clinical exploration of NEUK203-13 Injection in patients with advanced small cell lung cancer or other neuroendocrine tumors(NETs). Its primary focus is on safety, while simultaneously gathering preliminary signals on whether the therapy can control tumors, thereby laying the foundation for subsequent clinical development.

DETAILED DESCRIPTION:
NEUK203-13 Injection is a chimeric antigen receptor (CAR)-natural killer (NK) cell therapy (CAR-NK) derived from induced pluripotent stem cells (iPSCs). Through site-specific gene editing, it expresses a CAR structure targeting Delta-like Protein 3 (DLL3). Specifically, the CAR construct is introduced into NK cells via transgenic engineering, enabling precise recognition and elimination of malignant/cancer cells expressing the specific antigen DLL3. Beyond CAR molecular transgenesis, an IL-15RF fusion gene is inserted at the CD38 locus to enhance the pharmacokinetic (PK) properties of CAR-iNK cells. Additionally, the immune checkpoint receptor TIM3 is knocked out to improve resistance to the immunosuppressive tumor microenvironment, and a variant CD16 (vCD16, a cleavage-resistant CD16) is inserted to augment antibody-dependent cellular cytotoxicity (ADCC) when used in combination with therapeutic antibodies.

Using clinical-scale production batches and processes, in vitro pharmacodynamic studies and evaluations of NEUK203-13 Injection were conducted across multiple dimensions, including:

1. Nonspecific cytotoxicity against target cells (human chronic myelogenous leukemia cell line K562) at different process stages and in fresh bulk cells;
2. Specific cytotoxicity against tumor cells (small cell lung cancer cell lines SHP-77 and H82 with high DLL3 expression, and the human B-lymphoblastic leukemia cell line NALM6-DLL3 with stable exogenous DLL3 expression as target cells);
3. Cell viability post cryopreservation and thawing;
4. Cytotoxic activity (both nonspecific and specific) post cryopreservation and thawing.

NEUK203-13 represents an iterative upgrade of the first-generation product NEUK200-13. The accelerated advancement of NEUK203-13 into clinical research is based on the established clinical safety data of NEUK200-13 and the superior preclinical data of NEUK203-13.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understand and voluntarily sign the Informed Consent Form (ICF);
* 2. Aged ≥ 18 years and < 75 years at the time of signing the ICF, regardless of gender;
* 3. Pathologically confirmed neuroendocrine tumors, including small cell lung cancer (SCLC), etc.;
* 4. Previous failure or intolerance to systemic therapy, or recurrence after remission: among them, patients with small cell lung cancer must have received at least platinum-based chemotherapy with or without PD-1/PD-L1 inhibitors in previous treatments, with imaging evidence of disease progression after treatment;
* 5. Must provide tissue samples for biomarker analysis, preferably newly obtained tissues. For patients unable to provide newly obtained tissues, 4 unstained sections of archived formalin-fixed, paraffin-embedded (FFPE) tissues can be provided (at least 1 patient with high DLL3 expression shall be enrolled in each dose group: high expression is defined as positive staining in ≥ 50% of tumor cells; preference is given to enrolling DLL3-positive patients);
* 6. Have at least one measurable lesion as the target lesion (per RECIST v1.1 criteria);
* 7. Expected survival ≥ 3 months;
* 8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* 9. Have adequate bone marrow reserve and organ function within 7 days before the first administration of NEUK203-13 Injection:
* 10. Sufficient bone marrow function (no supportive therapy within 14 days before the first administration): hemoglobin (Hb) ≥ 90 g/L, platelets (PLT) ≥ 75 × 10⁹/L, absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
* 11. Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN), total bilirubin (TBIL) < 1.5 × ULN;
* 12. Renal function: serum creatinine (Scr) ≤ 1.5 × ULN and creatinine clearance rate (Ccr) ≥ 60 mL/min (calculated according to the Cockcroft-Gault formula); Coagulation function: prothrombin time (PT) ≤ 1.5 × ULN, international normalized ratio (INR) ≤ 2.0;
* 13. Female patients of childbearing potential or male patients whose partners are of childbearing potential agree to use highly effective contraceptive measures from any dose administration in the study until 6 months after the last dose of the study.

Exclusion Criteria:

* 1. Mixed carcinoma with non-neuroendocrine tumor components;
* 2. Active brain metastases (patients with stable disease for 3 months after treatment without the need for continued glucocorticoid therapy are eligible for enrollment); known leptomeningeal metastases; isolated central nervous system (CNS) disease progression without evidence of progression outside the CNS;
* 3. A history of hypersensitivity to interleukin-2 (IL-2), fludarabine, cyclophosphamide, tocilizumab, or any component of the infusion product formulation; or patients with a history of specific allergic disorders (asthma, rubella, eczematous dermatitis);
* 4. Prior receipt of any of the following treatments:
* 5. Any systemic antineoplastic therapy within 4 weeks or 5 half-lives prior to the first administration of NEUK203-13 Injection, whichever is shorter;
* 6. Radiotherapy not involving the thoracic cavity within 2 weeks prior to the first administration of NEUK203-13 Injection, or radiotherapy involving the thoracic cavity within 4 weeks prior to the first administration of the study drug, whichever is longer;
* 7. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study;
* 8. Prior vaccination with an antineoplastic vaccine, or receipt of a live vaccine within 4 weeks prior to the first administration of NEUK203-13 Injection;
* 9. Major surgery or severe trauma within 4 weeks prior to the first administration of NEUK203-13 Injection;
* 10. Failure of toxicities from prior antineoplastic therapy to resolve to ≤ Grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) (except alopecia) or to the level specified in the inclusion/exclusion criteria, whichever is more stringent;
* 11. Active autoimmune disease or a history of autoimmune disease (e.g., interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); exceptions include patients with vitiligo, patients with a history of childhood asthma/allergies that have resolved completely and require no intervention in adulthood, patients with autoimmune-mediated hypothyroidism receiving a stable dose of thyroid replacement hormone, and patients with type 1 diabetes receiving a stable dose of insulin;
* 12. A history of immunodeficiency, including positive HIV test results, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation;
* 13. Severe infection (CTCAE > Grade 2) within 4 weeks prior to the first administration of NEUK203-13 Injection, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; baseline chest imaging indicating active pulmonary inflammation; or presence of signs and symptoms of infection requiring oral or intravenous antibiotic therapy within 2 weeks prior to the first administration of the study drug (except for prophylactic antibiotic use);
* 14. Tuberculosis infection identified by medical history or CT examination; Active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (positive anti-HCV antibodies and HCV-RNA above the lower limit of detection of the assay), or positive syphilis test results (including positive RPR or TPPA);
* 15. Prior diagnosis of any other malignant tumor, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or breast cancer, or adequately treated localized prostate cancer;
* 16. Pregnant or lactating women;
* 17. Uncontrolled concurrent diseases, including but not limited to: documented cerebrovascular events (stroke or transient ischemic attack) within 6 months prior to the first administration of the study drug, symptomatic congestive heart failure, left ventricular ejection fraction (LVEF) < 50%, uncontrolled hypertension, unstable angina pectoris, uncontrolled arrhythmias, severe chronic gastrointestinal disease with diarrhea, or severe dyspnea requiring oxygen therapy;
* 18. A definite history of neurological or psychiatric disorders that, in the investigator's judgment, may affect the patient's cognitive function or compliance, including unstable epilepsy, dementia, schizophrenia, etc.; or psychiatric illnesses/social conditions that may affect study compliance, significantly increase the risk of adverse events, or impair the patient's ability to provide written informed consent;
* 19. Other factors judged by the investigator that may force the patient to terminate the study prematurely, such as severely abnormal laboratory test results, and/or family or social factors that may affect patient safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of Adverse Events (AEs) / Serious Adverse Events (SAEs) / Adverse Events of Special Interest (AESIs). | 12 months
  This endpoint aims to systematically monitor, record, and evaluate the safety profile of the study treatment by assessing the incidence, severity, duration, and causal relationship of Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) throughout the study period.

SECONDARY OUTCOMES:
Detect the number of NEUK203-13 cells in peripheral blood and calculate the PK parameters. | 12 months
  Quantification of NEUK203-13 Cells in Peripheral Blood and Pharmacokinetic (PK) Parameter Calculation
Ratio of DLL3 expression in tumor tissues versus response rate | 12 months
  Correlation Analysis Between DLL3 Expression Ratio in Tumor Tissues and Clinical Response Rate
Objective Response Rate (ORR) | 12 months
  The proportion of evaluable patients who achieve a complete response (CR) or partial response (PR) confirmed by two consecutive assessments separated by a minimum 4-week interval. CR is defined as the disappearance of all target and non-target lesions with no new lesions detected; PR refers to a ≥30% reduction in the sum of the longest diameters of target lesions, with no progression of non-target lesions or new lesions. ORR will be calculated as the percentage of patients with CR or PR relative to the total evaluable study cohort.
Duration of Response (DoR) | 12 months
  The time interval from the first documentation of CR or PR (per the above criteria) to the first confirmed occurrence of disease progression (per RECIST v1.1) or death from any cause, whichever occurs first. For patients who maintain a response until the end of the study, DoR will be censored at the date of the last tumor assessment.
Disease Control Rate (DCR) | 12 months
  The percentage of evaluable patients whose disease is controlled, encompassing those with CR, PR, and stable disease (SD). SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, with the sum of target lesion diameters changing by <30% (increase) and <20% (decrease) from baseline. DCR will be calculated as the proportion of patients with CR, PR, or SD relative to the total evaluable cohort, with SD required to last for a minimum of the predefined assessment cycle to be included.

OTHER OUTCOMES:
Detect the cytokines associated with the tumor cell killing process (IFN-γ, TNF-α) in peripheral blood. | 12 months
  The absolute concentration of IFN-γ and TNF-α in peripheral blood at each time point; The dynamic changes in cytokine levels relative to baseline values (calculated as percentage change or fold change); The correlation between cytokine level fluctuations and clinical endpoints (e.g., objective response rate, disease control rate) or biomarker changes (e.g., tumor cell burden, immune cell subsets).

CONTACTS AND LOCATIONS:
Overall Officials: Shuhang Wang, PhD, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital of CICAMS, Beijing, China

IPD SHARING:
Plan to Share IPD: No